CLINICAL TRIAL: NCT05089032
Title: The Practice of Providing Palliative Care in the Situation of the COVID-19 Pandemic in the Perspective of Physicians and Nurses - Survey Study (PEOpLe-C19-EN Study)
Brief Title: The Practice of Providing Palliative Care in the Situation of the COVID-19 Pandemic
Acronym: PEOpLeC19-EN
Status: Completed | Type: Observational
Sponsor: Masaryk University (Other)
Collaborators: European Society of Intensive Care Medicine (Other); European Society of Anaesthesiology and Intensive Care (Other); Brno University Hospital (Other)
Responsible Party: Principal Investigator, Jan Malaska, Head of research group, Masaryk University
Other Study IDs: PEOpLe-C19-EN
Record Dates: First submitted 2021-10-21; First posted 2021-10-22 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: COVID-19 Pandemic; End-of-life
Keywords: covid-19; Palliative Care; end-of-life
MeSH Terms: conditions — COVID-19; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Physicians
- Nurses

SUMMARY:
The practice of providing palliative care in the situation of the COVID-19 pandemic in the perspective of physicians and nurses - survey study (PEOpLe-C19 study)

DETAILED DESCRIPTION:
Pandemic of coronavirus SARS-CoV-2 (Severe Acute Respiratory Syndrome coronavirus 2) causing the disease COVID-19 (Coronavirus Disease 2019) overwhelmed healthcare and brought new challenges and stressful situations. In a short time, intensive care units (ICU) capacities were filled in many countries and regions. Due to the need for an excessive number of patients requiring intensive care, physicians and nurses who do not routinely provide care to critically ill patients or do not have the appropriate training (non-ICU clinician) were involved in the care of COVID-19 patients. In this context, ICU directly dedicated to caring for patients with COVID-19 ARDS (Acute Respiratory Distress Syndrome) was also opened. Non-ICU clinicians were more or less involved together with the standard ICU staff in palliative care, including End-of-Life decision (EOLD) making, even in a situation of limited, scarce resources (equipment or personnel). New workplace and scope of work, which did not correspond to the standard activity or education, most likely led to an increased stress load. EOLD can also be one of the factors leading to increased stress levels. The project aims to describe the practice of palliative care for patients with COVID-19 in a situation of pandemic COVID-19 and to identify factors leading to possible moral distress related to EOLD.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare providers (physicians/nurses)
* Involvement in care for patients with COVID-19 admitted at intensive care unit

Exclusion Criteria:

* Non-ICU staff
* not involved in care for patients with COVID-19

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Healthcare providers (physicians and nurses) providing care to patients with COVID-19 admitted at ICU in period of COVID-19 pandemic.
Sampling Method: Non-Probability Sample
Enrollment: 215 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-02-29 (Actual); Study Completion 2024-02-29 (Actual)

PRIMARY OUTCOMES:
Change of practice of providing palliative care at ICU in COVID-19 pandemic | Through study completion, an average of 1 month
  Change of practice of providing palliative care including EOLD practice in patients with COVID-19 admitted at ICU during pandemic.

SECONDARY OUTCOMES:
Identify factors leading to moral distress during the COVID-19 pandemic | Through study completion, an average of 1 month
  Identify factors leading to moral distress during COVID-19 pandemic and describe possible different risk factors by profession

CONTACTS AND LOCATIONS:
Overall Officials: Tereza Prokopova, MD, Principal Investigator — University Hospital Brno
Locations (1):
- Masaryk University, Brno, Czechia

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2021-06-15): https://cdn.clinicaltrials.gov/large-docs/32/NCT05089032/Prot_000.pdf